CLINICAL TRIAL: NCT06691997
Title: The Impact of Glycemic Control on Rheumatoid Arthritis Disease Activity in Diabetic Patients
Brief Title: The Impact of Glycemic Control on Rheumatoid Arthritis Disease Activity on Diabetic Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Khedr Nady Abd Elaziz, Assistant lecture, Assiut University
Other Study IDs: DM and Rheumatoid Arthritis
Record Dates: First submitted 2024-10-27; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Rheumatoid Arthritis (RA; Diabetes Mellitus
Keywords: glycemic control
MeSH Terms: conditions — Arthritis, Rheumatoid; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group 1: RA patients with Type 2 diabetes

SUMMARY:
The incidence of DM is unclear in RA but most prior data suggest that DM or insulin resistance in RA has risen because of activation of the immune system and/or RA therapy .

Besides, RA causes joints to become stiff, swollen, and agonizing. As a result, the patient may not want to exercise or move. One study found that 42% of people with RA are not physically active. the aim of this study is To evaluate the glycemic status among RA patients with Type 2 diabetes and its association with disease activity.

DETAILED DESCRIPTION:
Taking the potential link between DM and RA into consideration, detection and control of DM will significantly increase prolonged prognosis and therefore decrease the economic burden of RA patients and death rate. The aim of this research is to examine diabetic RA's glycemic status and to assess the relationship between RA and DM's clinical characteristics as well as the therapy response in RA patients with diagnosed DM. Keeping an eye on glycemic control in RA patients could prevent metabolic and cardiovascular comorbidities in those susceptible patients.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic patients
* rheumatoid arthritis patients

Exclusion Criteria:

* gestional diabetes
* type 1 diabetic patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients above age of 18 years old diagnosed with Rheumatoid Arthritis and DM
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-12 (Estimated); Primary Completion 2026-11-14 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Fasting blood glucose | baseline
  correlation between type 2 diabetes control and rheumatoid arthritis activity

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed khedr Nady, Principal Investigator — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
According to result of search

REFERENCES:
- See also: Wasserman A. Rheumatoid Arthritis: Common Questions About Diagnosis and Management. Am Fam Physician. 2018 Apr 1;97(7):455-462. PMID: 29671563. — https://pubmed.ncbi.nlm.nih.gov/29671563/
- See also: Almutairi KB, Nossent JC, Preen DB, Keen HI, Inderjeeth CA. The Prevalence of Rheumatoid Arthritis: A Systematic Review of Population-based Studies. J Rheumatol. 2021 May;48(5):669-676. doi: 10.3899/jrheum.200367. Epub 2020 Oct 15. PMID: 33060323. — https://pubmed.ncbi.nlm.nih.gov/33060323/
- See also: Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Meas — https://pubmed.ncbi.nlm.nih.gov/20872595/
- See also: Schoels M, Knevel R, Aletaha D, Bijlsma JWJ, Breedveld FC, Boumpas DT, Burmester G, Combe B, Cutolo M, Dougados M, Emery P, van der Heijde D, Huizinga TWJ, Kalden J, Keystone EC, Kvien TK, Martin-Mola E, Montecucco C, de Wit M, Smolen JS. Evidence for tr — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3015093/
- See also: Jiang P, Li H, Li X. Diabetes mellitus risk factors in rheumatoid arthritis: a systematic review and meta-analysis. Clin Exp Rheumatol. 2015 Jan-Feb;33(1):115-21. Epub 2014 Dec 22. PMID: 25535750. — https://pubmed.ncbi.nlm.nih.gov/25535750/